CLINICAL TRIAL: NCT01093586
Title: Umbilical Cord Blood (UCB) Allogeneic Stem Cell Transplant for Hematologic Malignancies
Brief Title: Donor Umbilical Cord Blood Stem Cell Transplant in Treating Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3Z07; NCI-2009-01319 (Other: NCI/CTRP); CASE3Z07 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2010-03-24; First posted 2010-03-26 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Erythroleukemia (M6a); Adult Nasal Type Extranodal NK/T-cell Lymphoma; Adult Pure Erythroid Leukemia (M6b); B-cell Adult Acute Lymphoblastic Leukemia; B-cell Childhood Acute Lymphoblastic Leukemia; Blastic Phase Chronic Myelogenous Leukemia; Burkitt Lymphoma; Childhood Acute Erythroleukemia (M6); Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Megakaryocytic Leukemia (M7); Childhood Acute Minimally Differentiated Myeloid Leukemia (M0); Childhood Acute Monoblastic Leukemia (M5a); Childhood Acute Monocytic Leukemia (M5b); Childhood Acute Myeloid Leukemia in Remission; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Juvenile Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Previously Treated Myelodysplastic Syndromes; Prolymphocytic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Secondary Myelofibrosis; Splenic Marginal Zone Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia; T-cell Adult Acute Lymphoblastic Leukemia; T-cell Childhood Acute Lymphoblastic Leukemia; T-cell Large Granular Lymphocyte Leukemia; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Congenital Abnormalities; Leukemia, Erythroblastic, Acute; Lymphoma, Extranodal NK-T-Cell; Blast Crisis; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Juvenile; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Cytogenetic Analysis; In Situ Hybridization, Fluorescence; Busulfan; Cyclophosphamide; Antilymphocyte Serum; thymoglobulin; Methylprednisolone; Methylprednisolone Hemisuccinate; Methylprednisolone Acetate; Cyclosporine; Cyclosporins; Mycophenolic Acid; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): PREPARATIVE REGIMEN: Patients receive oral busulfan on days -8 to -5, cyclophosphamide IV on days -4 to -3, and anti-thymocyte globulin or methylprednisolone IV on days -3 to -1. TRANSPLANTATION: Patients undergo a double-unit umbilical cord blood allogeneic stem cell transplantation on day 0. GRAFT-VS-HOST DISEASE PROPHYLAXIS: Beginning on day -2, patients receive cyclosporine IV and taper beginning on day 100. Patients also receive mycophenolate mofetil IV or orally on days -3 to 45.
  Interventions: Procedure: double-unit umbilical cord blood transplantation; Other: cytogenetic analysis; Procedure: bone marrow aspiration; Other: fluorescence in situ hybridization; Drug: busulfan; Drug: cyclophosphamide; Drug: anti-thymocyte globulin; Drug: methylprednisolone; Drug: cyclosporine; Drug: mycophenolate mofetil; Other: flow cytometry; Procedure: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Procedure: double-unit umbilical cord blood transplantation — Undergo transplantation
Other: cytogenetic analysis — Correlative studies
Procedure: bone marrow aspiration — Correlative studies
Other: fluorescence in situ hybridization — Correlative studies
  Other Names: fluorescence in situ hybridization (FISH)
Drug: busulfan — Given orally
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon; Myelosan
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana; Enduxan
Drug: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Drug: methylprednisolone — Given IV
  Other Names: A-MethaPred; Depo-Medrol; Medrol; MePRDL; Solu-Medrol; Wyacort
Drug: cyclosporine — Given IV
  Other Names: 27-400; ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given orally or IV
  Other Names: Cellcept; MMF
Other: flow cytometry — Correlative studies
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo transplantation

SUMMARY:
RATIONALE: Giving chemotherapy before a donor umbilical cord blood transplant (UCBT) helps stop the growth of cancer and abnormal cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the stem cells from an unrelated donor, that do not exactly match the patient's blood, are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving antithymocyte globulin before transplant and cyclosporine and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well donor umbilical cord blood stem cell transplant works in treating patients with hematologic malignancies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To establish the day +180 overall survival after a myeloablative unrelated double unit UCBT in a single institution setting.

SECONDARY OBJECTIVES:

1. To determine the rates of hematologic and immune reconstitution in patients with high risk hematologic malignancies, who are undergoing myeloablative chemotherapy followed by infusion of double unit UCBT.
2. To determine the contribution of each umbilical cord unit to immune reconstitution with a focus on both initial (day +21 BM, and +28 PB) and sustained engraftment (day +100 BM; PB at +14, +21, +28, +35, +42, +60, +100, +180, +1 and 2 years).
3. To determine the probability of overall survival and disease free survival at one and two years.
4. To describe the incidence of disease recurrence at one and two years in patients post UCBT.
5. To describe the incidence of acute GVHD and chronic GVHD at 100 days and at one year, respectively.
6. To determine the incidence of day 100 and 180 treatment related mortality.
7. To determine the incidence of serious infectious complications in the first year after transplant.
8. To determine the incidence of donor-derived neutrophil and platelet recovery.
9. To determine the incidence of secondary lymphoproliferative diseases following transplantation with umbilical cord blood.

OUTLINE:

PREPARATIVE REGIMEN: Patients receive oral busulfan every 6 hours on days -8 to -5, cyclophosphamide IV on days -4 to -3, and anti-thymocyte globulin or methylprednisolone IV on days -3 to -1.

TRANSPLANTATION: Patients undergo double-unit umbilical cord blood allogeneic stem cell transplantation on day 0.

GRAFT-VS-HOST DISEASE PROPHYLAXIS: Beginning on day -2, patients receive cyclosporine IV and taper beginning on day 100. Patients also receive mycophenolate mofetil IV or orally every 8 hours on days -3 to 45. After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be diagnosed with one of the following hematological malignancies: acute myelogenous leukemia (AML), acute lymphoblastic leukemia, non-Hodgkin's lymphoma, myelodysplastic syndrome (MDS), chronic myelogenous leukemia (CML), and myeloproliferative and lymphoproliferative disorders
* AML--First remission (CR1) with high risk features including a known prior diagnosis of myelodysplasia (MDS); therapy related AML; white cell count at presentation > 100,000; presence of extramedullary leukemia at diagnosis; unfavorable AML subtype (M0, M5-M7); poor cytogenetic markers (abnormalities of chromosome 5, 7 or 8, 11q23, Philadelphia chromosome, complex karyotype)
* AML--Second remission (CR2) or subsequent remission
* AML--Relapse/Persistent Disease with < 20% bone marrow blasts
* ALL--First remission (CR1) at high risk for relapse as defined by: B cell ALL white blood cell count (WBC) at presentation > 30,000 (T cell ALL WBC > 100,000); presence of high-risk cytogenetic abnormality such as t(9;22), t(1;19), t(4;11) or other MLL rearrangements (11q23), t(8;14)
* ALL--Second remission (CR2) or subsequent remission
* ALL--Relapse/Persistent Disease with < 20% bone marrow blasts
* Non-Hodgkin Lymphoma--Induction failure or relapse and sensitive to most recent chemotherapy
* MDS--Low or Intermediate-1 International Prognostic Scoring System (IPSS) score with: life-threatening cytopenia(s); and/or red cell or platelet transfusion dependence
* MDS--ANC < 500, recurrent infections, PRBC transfusions > 2 units/month, poor risk cytogenetics, platelet transfusion dependence
* MDS--Intermediate-2 or High IPSS score
* CML--Chronic phase I (CP1) and resistant to or intolerant of tyrosine kinase inhibitors (i.e. imatinib, dasatinib, etc.)
* CML--CP2 or subsequent chronic phase, including chronic phase achieved after induction therapy for blast crisis
* Myeloproliferative and lymphoproliferative disorders--eligibility to be determined by a consensus of the physicians on the Case Comprehensive Cancer Center Leukemia/Lymphoma Multidisciplinary Committee
* Myeloproliferative and lymphoproliferative disorders--must have evidence of disease acceleration to be a candidate for umbilical cord blood transplant; myeloproliferative disorders eligible for transplant include chronic myelomonocytic leukemia (CMML) with high IPSS score and myelofibrosis
* Myeloproliferative and lymphoproliferative disorders--potential lymphoproliferative disorders eligible for transplant include chronic lymphocytic leukemia, prolymphocytic leukemia, and large granular lymphocytic leukemia
* Good performance status: Karnofsky >= 70 % or ECOG 0-1
* Calculated creatinine clearance >= 60 mL/min, or measured creatinine clearance >= 60 mL/min (by 24-hour urine collection) if creatinine >= 1.5 or history of renal dysfunction
* Hepatic Transaminases < 4 x upper limit normal (ULN); total bilirubin < 2.5 mg/dL, unless the patient has a history of benign congenital hyperbilirubinemia (Gilbert's syndrome)
* Normal cardiac function by echocardiogram or radionuclide scan, (left ventricular ejection fraction > 45%); if the left ventricular ejection fraction is between 40-50%, clearance by an adult cardiologist is required
* Pulmonary function tests demonstrating FEV1 > 60% of predicted for age
* Adults must have a DLCOva > 60% normal
* For patients unable to complete pulmonary function tests clearance by an adult pulmonologist is required
* Patients will be eligible for the clinical trial under the following conditions: they do NOT have an HLA-A/B/DR B1 identical RELATED bone marrow donor; they do NOT have a 6/6 HLA-identical matched unrelated adult donor; OR a matched related donor transplant is not in the best interest of the patient (i.e., patient's condition precludes waiting on the donor, too much time to prepare the donor, the donor is ineligible due to medical reasons, or in the case of high risk disease a related donor is not appropriated (syngeneic transplant); the decision must be agreed upon by the consensus of physicians on the Case Comprehensive Cancer Center Leukemia/Lymphoma Multidisciplinary Committee; OR their condition precludes waiting to search and find a donor in the National Marrow Donor Registry

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* HIV or HTLV-1 positivity
* Any leukemia with a morphologic relapse or persistent disease in the BM with >= 20% blasts (cytogenetic relapse without morphologic evidence of relapse, or cytogenetic persistent disease is acceptable)
* Active extramedullary leukemia, including CNS disease
* Prior hematopoietic stem cell transplant (autologous or allogeneic)
* Uncontrolled infection
* Patient has an identical related bone marrow donor or a 6/6 HLA-identical matched unrelated donor
* Any patient who is unable to provide informed consent or comply with the requirements of the protocol

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2007-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Cooper, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from medical hospital from 9/2007 thru 2/2013.
Period: Overall Study
Arm/Group | Arm I
Started | 14
Completed | 11
Not Completed | 3
Not completed — Failed to engraft | 3

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 14
Age, Customized [Count of Participants; unit: Participants]
  10-19 yrs | 2
  20-29 yrs | 2
  30-39 yrs | 3
  40-49 yrs | 5
  50-59 yrs | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Number of participants alive at 180 days post engraftment.
Time Frame: On day +180
Population: All participants that went on study, whether completing engraftment or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants | 8

2. Secondary Outcome: Hematologic Engraftment
Description: Number of participants that were able to complete engraftment by day 42.
Time Frame: On day +42
Population: Participants that went on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants | 10

3. Secondary Outcome: Overall Survival
Description: Number of participants that were alive.
Time Frame: At 1 year
Population: Participants that completed engraftment. 10 participants completed engraftment by day 42 and 1 participant completed engraftment by day 46.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 11
Participants | 6

4. Secondary Outcome: Overall Survival
Description: Number of participants that were alive.
Time Frame: At 2 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 11
Participants | 4

5. Secondary Outcome: Disease Free
Description: Number of participants that were disease free
Time Frame: At 1 year
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 11
Participants | 4

6. Secondary Outcome: Disease Free
Description: Number of participants that were disease free
Time Frame: At 2 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 11
Participants | 4

7. Secondary Outcome: Recurrence or Relapse
Description: Number of subjects that had disease recurrence
Time Frame: one year in patients post UCBT
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 11
Participants | 2

8. Secondary Outcome: Recurrence or Relapse
Description: Number of subjects that had disease recurrence
Time Frame: two years post transplant
Population: Subjects who had completed engraftment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 11
Participants | 2

9. Secondary Outcome: Transplant Related Mortality
Description: Number of subjects that died because of transplant
Time Frame: On day 100 post transplant
Population: Participants that went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants | 2

10. Secondary Outcome: Transplant Related Mortality
Description: Number of subjects that died because of transplant
Time Frame: On day 180 post transplant
Population: All participants that went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants | 6

11. Secondary Outcome: Occurrence of Serious Infections
Description: Number of participants that had infections
Time Frame: 1 year
Population: All participants that went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants | 13

12. Secondary Outcome: Immune Reconstitution
Description: Immunodificency panel to see recovery of immune system. Number of participants that recovered.
Time Frame: Periodically for 2 years
Population: Data not collected, panel not done because of funding.
Arm/Group | Arm I
Number analyzed (Participants) | 0

13. Secondary Outcome: Toxicity Related to UCB Transplantation and Cytoreduction as Assessed by CTC v3.0
Description: Number of participants that experienced toxicity related to the transplant
Time Frame: by day +42
Population: Patients that received transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 11
Participants | 8

14. Secondary Outcome: Incidence of Acute Graft-versus-host Disease (GVHD)
Description: Number of participants that had acute GVHD
Time Frame: At 100 days
Population: All participants who went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants | 11

15. Secondary Outcome: Incidence of Chronic GVHD
Description: Number of participants that have chronic GVHD. Chronic GVHD will be diagnosed and graded on clinical and histological criteria from the Center for International Blood and Marrow Transplant Research (CIBMTR)
Time Frame: At 1 year
Population: All participants that went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I
Number analyzed (Participants) | 14
Participants | 1

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from participant start on study to going off study up to a period of 2 years.
Description: Non serious events were not collected. The protocol was assessing efficacy of cord blood in transplants, therefore the research was only gathering SAEs of grade 3 or 4.
Arm/Group | Arm I
All-Cause Mortality (participants affected / at risk) | 11/14
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=14)
Diarrhea (Gastrointestinal disorders) | 3 (4)
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 1 (1)
Death not associated with CTCAE term - Multi-organ failure (General disorders) | 3 (3)
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Death not associated with CTCAE term - Death NOS (General disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
Bone marrow cellularity - Primary graft failure (Blood and lymphatic system disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Product Issues) | 2 (2) — Catheter related
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Brain (encephalitis, infectious) (Nervous system disorders) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes